CLINICAL TRIAL: NCT04435951
Title: The Effect Of Temporomandibular Joint Dysfunction On Pain, Quality Of Life And Psychological Status
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Tolgahan YILDIZ, Research Assistant, Hacettepe University
Other Study IDs: Hacettepe FTR
Record Dates: First submitted 2020-06-05; First posted 2020-06-17 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Temporomandibular Joint Dysfunction
Keywords: Temporomandibular joint; Dysfunction; Pain; Quality of life
MeSH Terms: conditions — Temporomandibular Joint Disorders; Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 (with TMJD): Group 1, consists of 60 patients diagnosed with Temporomandibular Joint Dysfunction (TMJD) according to the Research Diagnostic Criteria for Temporomandibular Disorders by a specialist and experienced dentist in TMJD.
  Interventions: Other: Evaluation
- Group 2 (without TMJD): Group 2, consists of 60 individuals who did not exhibit TMJD symptoms and have not TMJD diagnosis.
  Interventions: Other: Evaluation

INTERVENTIONS:
Other: Evaluation — No attempt was made to the individuals in Group 1 and Group 2. Individuals were only evaluated.

SUMMARY:
The aim of this study was to investigate the effects of temporomandibular joint dysfunction (TMJD) on pain, quality of life and psychological status.

A total of one hundred twenty people participated in the study, sixty with TMJD symptoms (according to the Research Diagnostic Criteria for Temporomandibular Disorders) and sixty without TMJD symptoms. The severity of temporomandibular joint (TMJ) pain and headache was assessed using a visual analog scale (VAS), pain threshold using an algometer, anxiety and depression levels with the Hospital Anxiety and Depression Scale (HADS), and the quality of life level was assessed by Short Form-36 (SF-36).

Treatment of TMJD with appropriate therapies and psychological support techniques may reduce TMJD symptoms and improve patients' quality of life and psychological status.

DETAILED DESCRIPTION:
Temporomandibular joint dysfunction (TMJD) occurs as a result of the impaired functioning of the structures of the masticatory system. This disruption affects the chewing muscles, temporomandibular joint (TMJ), and related structures around the joint. TMJD can produce signs and symptoms, including pain in the TMJ and chewing muscles, restricted mouth opening, and articular sounds such as clicking and/or crepitus. Other symptoms include TMJ pain, limitation in joint movements, difficulty in chewing, jaw locking (trismus), lateral deviation of the jaw, tenderness in the TMJ and chewing muscles, tinnitus and pain, dizziness, and head and neck pain.

However, to the best of the investigator's knowledge, no previous studies have examined the relationship between quality of life, pain, and psychological status in individuals with TMJD. This study was designed to investigate whether a relationship between pain, quality of life, and psychological status in individuals with TMJD and asymptomatic individuals without TMJD.

One hundred twenty individuals were included in this study performed between March and July 2017 at the Gazi University and Ankara Yıldırım Beyazıt University Dentistry Faculties, Turkey. The research was designed as a controlled, observational, cross-sectional study. Sixty of the 165 individuals presenting with TMJD symptoms were diagnosed with TMJD by a specialist dentist, and those meeting the inclusion criteria were enrolled in the first group. Sixty individuals who met the inclusion criteria out of 143 individuals who did not exhibit TMJD symptoms were enrolled in the second group. These two groups were established based on clinical and radiological examination results. TMJD was diagnosed by professional and experienced dentists using the Research Diagnostic Criteria for Temporomandibular Disorders (RDC/TMD). RDC/TMD has been described as the gold standard physical examination method in the clinical diagnosis of TMD.

Individuals agreeing to take part in the study were included after signing informed consent forms. Ethical committee permission was granted by the Ankara Yıldırım Beyazıt University Social and Humanities Ethics Committee (date: 02.08.2016, no: 356).

Individuals who were able to understand and speak Turkish and cooperate, and aged 17 years or older were included in the study.

Inclusion criteria for Group 1 were articular sounds in the form of clicks or crepitation from the TMJ during mouth opening or chewing, sensitivity and pain in the TMJ at palpation, no treatment for the TMJ in the previous six months, and presence of TMJD symptoms for at least three months. Inclusion criteria for Group 2, maximum mouth opening exceeding 30 mm, absence of articular sounds such as TMJ click or crepitation during mouth opening and closing and/or chewing activity, and absence of tenderness and pain in the TMJ and chewing muscles at palpation.

Exclusion criteria for Group 1 were the absence of at least one of the TMJD symptoms, absence of diagnosis of TMJD and the presence of a history of tumor, cervical discopathy, orthopedic and rheumatic pathologies, head, neck and/or jaw surgery and pregnancy.

Exclusion criteria for Group 2 were the presence of at least one of the symptoms of TMJD, the presence of a history of tumor, cervical discopathy, orthopedic and rheumatic pathologies, head, neck and/or jaw surgery, and pregnancy.

G * Power (V.3.1.9.2, Germany) software was used to calculate the sample size. Analyses were performed to investigate significant differences in the pressure pain threshold (PTT), quality of life, and psychological evaluation results between the groups (α = 0.05 and β = 0.20). The analysis showed that at least 19 individuals in each group and at least 38 individuals in total would be sufficient.

Socio-demographic (age, sex, height, weight, educational status) and clinical data (history of bruxism, dominant side, side of the problem, duration of symptoms, dominant chewing side, sleeping position, tinnitus/pain, chewing difficulty, and parafunctional oral habits status) of individuals meeting the inclusion criteria were recorded onto an evaluation form.

Individuals in both groups were asked to mark TMJ pain and headache on a 10 cm straight line using a visual analog scale (VAS), and the results were recorded in cm. Patients were asked about pain in bilateral resting and mobile positions of the TMJ. On the VAS scale, "0" indicates no pain, and "10" the most severe pain possible.

Muscle sensitivity was measured using an algometer (Baseline® dolorimeter/algometer, Pain Diagnosis, and Treatment Inc., Great Neck, NY, USA). The algometer is pressed gradually to the area where the sensitivity is to be measured, and the measurement is terminated as soon as the subject experiences pain. The PPTs of the anterior part of the temporalis muscle, the TMJ lateral capsule, and the masseter muscle were measured in the present study. Measurements were performed three times at 30-second intervals on both right and left sides. The mean values of the three measurements were recorded. PPT is defined as the lowest pressure force required to be applied to the tissue for the pain to occur. Results are expressed as kg/cm2.

The Hospital Anxiety and Depression Scale (HADS) was used to measure participants' anxiety and depression levels. The HADS scale was developed by Zigmond and Snaith and contains 14, with two sub-scales, one of seven questions (odd numbers) measuring anxiety, and another of seven questions (even numbers) measuring depression. Aydemir et al. conducted the Turkish validity and reliability study of HADS. Each question is scored between 0 and 3. The lowest possible scores for the depression and anxiety subscales were 0, and the maximum possible scores were 21. Subjects' depression and anxiety status are evaluated as normal/no symptoms (0-7 points), borderline abnormal/suspicious (8-10 points), and abnormal/definite (11-21 points), depending on the scores obtained.

Short Form-36 (SF-36) was used to assess the quality of life. Ware et al. developed the SF-36 in 1987 to determine overall health-related life quality. The scale consists of 36 questions and evaluates life quality in the previous four weeks in eight subscales and two main components. The subscales are; Physical Function (PF), Role Difficulty-Physical (RP), Body Pain (BP), General Health (GH), Vitality (V), Social Function (SF), Role Difficulty-Emotional (RE), and Mental Health (MH), while the main components are Physical Component Score (PCS) and Mental Component Score (MCS). The eight subscales assess health from 0 to 100 points. "0" indicates that health-related quality of life is poor, and 100 indicates the best possible quality of life, so higher scores indicate better quality of life. SF-36 was translated into Turkish by Koçyiğit et al. and has been subjected to validity and reliability studies.

The distributions of continuous variables such as age, body mass index (BMI), and SF-36 scores were examined using the Shapiro-Wilk test and normality graphs. Mean ± standard deviation (mean ± sd) and median (min-max: minimum-maximum) were used to express all continuous variables, while results for categorical variables such as gender and occupation were expressed as percentages (%). The independent samples t-test and Mann-Whitney U test were applied to determine the distribution of continuous variables such as SF-36 and HADS scores between groups 1 and 2. The relationship between the scale scores and pain threshold and pain severity was analyzed using Pearson and Spearman correlation analysis. The consistency of responses to SF-36 and HADS was examined using Cronbach's alpha coefficient. Statistical significance was set at p <0.05. All statistical analyses and calculations were performed on IBM SPSS Statistics 21.0 software (IBM Corp. Released 2012. IBM SPSS Statistics for Windows, Armonk, NY: IBM Corp., USA).

ELIGIBILITY:
Inclusion Criteria:

For Group 1 (group with TMJD):

* Patients diagnosed with TMJD
* Able to understand and speak Turkish and cooperate
* Aged 17 years or older and 65 years or younger
* Patients have articular sounds in the form of clicks or crepitation from the TMJ during mouth opening or chewing
* Sensitivity and pain in the TMJ at palpation
* Not receiving TMJ treatment in the past six months
* Presence of TMJD symptoms for at least three months For Group 2 (group without TMJD)
* Able to understand and speak Turkish and cooperate
* Aged 17 years or aged 17 years or older and 65 years or younger
* Maximum mouth opening 30 mm or more
* Absence of articular sounds such as TMJ click or crepitation during mouth opening and closing and/or chewing activity.
* Absence of tenderness and pain in the TMJ and chewing muscles at palpation

Exclusion Criteria:

For Group 1 (group with TMJD):

* Absence of at least one of the TMJD symptoms
* Presence of a history of tumor, cervical discopathy, orthopedic and rheumatic pathologies, head, neck and/or jaw surgery and pregnancy For Group 2 (group without TMJD)
* Presence of at least one of the symptoms of TMJD
* Presence of a history of tumor, cervical discopathy, orthopedic and rheumatic pathologies, head, neck and/or jaw surgery and pregnancy

Ages: 17 Years to 57 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Group 1 (60 patients, group with TMJD) consists of patients diagnosed with TMJD according to the Research Diagnostic Criteria for Temporomandibular Disorders by a specialist and experienced dentist in TMJD.
  Group 2 (60 healthy individuals, group without TMJD) consists of individuals who are evaluated by a specialist and experienced dentist in TMJD and who do not show symptoms of TMJD.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2017-07-24 (Actual); Study Completion 2020-05-25 (Actual)

PRIMARY OUTCOMES:
Temporomandibular joint pain severity and headache severity | 5 months
  Individuals in both groups were asked to mark TMJ pain and headache on a 10 cm straight line using a visual analogue scale (VAS), and the results were recorded in cm. Patients were asked about pain in bilateral resting and mobile positions of the TMJ. On the VAS scale, "0" indicates no pain, and "10" the most severe pain possible.

SECONDARY OUTCOMES:
Psychological status (anxiety and depression levels) | 5 months
  The Hospital Anxiety and Depression Scale (HADS) was used to measure participants' anxiety and depression levels. Each question was scored between 0 and 3. The lowest possible scores for the depression and anxiety subscales were 0, and the maximum possible scores were 21. Subjects' depression and anxiety status was evaluated as normal/no symptoms (0-7 points), borderline abnormal/suspicious (8-10 points) and abnormal/definite (11-21 points), depending on the scores obtained.
Short Form-36 | 5 months
  Short Form-36 (SF-36) was used to assess health-related quality of life. The scale consists of 36 questions and evaluates life quality in the previous four weeks in eight subscales and two main components. The eight subscales assess health from 0 to 100 points. "0" indicates that health-related quality of life is poor, and 100 indicates the best possible quality of life, so higher scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Nazım Tolgahan YILDIZ, MSc, Principal Investigator — Hacettepe University; Bahar KÜLÜNKOĞLU, PhD, Principal Investigator — Ankara Yildirim Beyazıt University
Locations (1):
- Ankara Yıldırım Beyazıt University Faculty of Health Sciences Department of Physiotherapy and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vedolin GM, Lobato VV, Conti PC, Lauris JR. The impact of stress and anxiety on the pressure pain threshold of myofascial pain patients. J Oral Rehabil. 2009 May;36(5):313-21. doi: 10.1111/j.1365-2842.2008.01932.x. Epub 2009 Feb 6. PMID 19210679
- [Result] Barbosa Tde S, Miyakoda LS, Pocztaruk Rde L, Rocha CP, Gaviao MB. Temporomandibular disorders and bruxism in childhood and adolescence: review of the literature. Int J Pediatr Otorhinolaryngol. 2008 Mar;72(3):299-314. doi: 10.1016/j.ijporl.2007.11.006. Epub 2008 Jan 3. PMID 18180045
- [Result] Chisnoiu AM, Picos AM, Popa S, Chisnoiu PD, Lascu L, Picos A, Chisnoiu R. Factors involved in the etiology of temporomandibular disorders - a literature review. Clujul Med. 2015;88(4):473-8. doi: 10.15386/cjmed-485. Epub 2015 Nov 15. PMID 26732121
- [Result] Suvinen TI, Hanes KR, Gerschman JA, Reade PC. Psychophysical subtypes of temporomandibular disorders. J Orofac Pain. 1997 Summer;11(3):200-5. PMID 9610309
- [Result] Wright AR, Gatchel RJ, Wildenstein L, Riggs R, Buschang P, Ellis E 3rd. Biopsychosocial differences between high-risk and low-risk patients with acute TMD-related pain. J Am Dent Assoc. 2004 Apr;135(4):474-83. doi: 10.14219/jada.archive.2004.0213. PMID 15127871
- [Result] Suvinen TI, Reade PC, Kemppainen P, Kononen M, Dworkin SF. Review of aetiological concepts of temporomandibular pain disorders: towards a biopsychosocial model for integration of physical disorder factors with psychological and psychosocial illness impact factors. Eur J Pain. 2005 Dec;9(6):613-33. doi: 10.1016/j.ejpain.2005.01.012. PMID 15978854
- [Result] Gameiro GH, da Silva Andrade A, Nouer DF, Ferraz de Arruda Veiga MC. How may stressful experiences contribute to the development of temporomandibular disorders? Clin Oral Investig. 2006 Dec;10(4):261-8. doi: 10.1007/s00784-006-0064-1. Epub 2006 Aug 22. PMID 16924558
- [Result] Krogstad BS, Jokstad A, Dahl BL, Vassend O. Relationships between risk factors and treatment outcome in a group of patients with temporomandibular disorders. J Orofac Pain. 1996 Winter;10(1):48-53. PMID 8995916
- [Result] Rocha CO, Peixoto RF, Resende CM, Alves AC, Oliveira AG, Barbosa GA. Psychosocial aspects and temporomandibular disorders in dental students. Quintessence Int. 2017;48(3):241-249. doi: 10.3290/j.qi.a37128. PMID 27834414
- [Result] Dahlstrom L, Carlsson GE. Temporomandibular disorders and oral health-related quality of life. A systematic review. Acta Odontol Scand. 2010 Mar;68(2):80-5. doi: 10.3109/00016350903431118. PMID 20141363
- [Result] Schierz O, John MT, Reissmann DR, Mehrstedt M, Szentpetery A. Comparison of perceived oral health in patients with temporomandibular disorders and dental anxiety using oral health-related quality of life profiles. Qual Life Res. 2008 Aug;17(6):857-66. doi: 10.1007/s11136-008-9360-3. Epub 2008 Jun 4. PMID 18523867
- [Result] Barros Vde M, Seraidarian PI, Cortes MI, de Paula LV. The impact of orofacial pain on the quality of life of patients with temporomandibular disorder. J Orofac Pain. 2009 Winter;23(1):28-37. PMID 19264033
- [Result] Bair MJ, Wu J, Damush TM, Sutherland JM, Kroenke K. Association of depression and anxiety alone and in combination with chronic musculoskeletal pain in primary care patients. Psychosom Med. 2008 Oct;70(8):890-7. doi: 10.1097/PSY.0b013e318185c510. Epub 2008 Sep 16. PMID 18799425
- [Result] Silva AA Jr, Brandao KV, Faleiros BE, Tavares RM, Lara RP, Januzzi E, Carvalho AB, Carvalho EM, Gomes JB, Leite FM, Alves BM, Gomez RS, Teixeira AL. Temporo-mandibular disorders are an important comorbidity of migraine and may be clinically difficult to distinguish them from tension-type headache. Arq Neuropsiquiatr. 2014 Feb;72(2):99-103. doi: 10.1590/0004-282X20130221. PMID 24604361
- [Result] Oliveira LK, Almeida Gde A, Lelis ER, Tavares M, Fernandes Neto AJ. Temporomandibular disorder and anxiety, quality of sleep, and quality of life in nursing professionals. Braz Oral Res. 2015;29:S1806-83242015000100265. doi: 10.1590/1807-3107BOR-2015.vol29.0070. PMID 26039910
- [Result] Dworkin SF, LeResche L. Research diagnostic criteria for temporomandibular disorders: review, criteria, examinations and specifications, critique. J Craniomandib Disord. 1992 Fall;6(4):301-55. No abstract available. PMID 1298767
- [Result] Schiffman E, Ohrbach R, Truelove E, Look J, Anderson G, Goulet JP, List T, Svensson P, Gonzalez Y, Lobbezoo F, Michelotti A, Brooks SL, Ceusters W, Drangsholt M, Ettlin D, Gaul C, Goldberg LJ, Haythornthwaite JA, Hollender L, Jensen R, John MT, De Laat A, de Leeuw R, Maixner W, van der Meulen M, Murray GM, Nixdorf DR, Palla S, Petersson A, Pionchon P, Smith B, Visscher CM, Zakrzewska J, Dworkin SF; International RDC/TMD Consortium Network, International association for Dental Research; Orofacial Pain Special Interest Group, International Association for the Study of Pain. Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) for Clinical and Research Applications: recommendations of the International RDC/TMD Consortium Network* and Orofacial Pain Special Interest Groupdagger. J Oral Facial Pain Headache. 2014 Winter;28(1):6-27. doi: 10.11607/jop.1151. PMID 24482784
- [Result] Daher, CRDM., Cunha, LFD., Ferreira, APDL., Souza, AISDO., Rêgo, TAM., Araújo, M. DGRD., & Silva, HJD. Pain threshold, sleep quality and anxiety levels in individuals with temporomandibular disorders. Revista CEFAC. 2018; 20(4); 450-458.
- [Result] Wewers ME, Lowe NK. A critical review of visual analogue scales in the measurement of clinical phenomena. Res Nurs Health. 1990 Aug;13(4):227-36. doi: 10.1002/nur.4770130405. PMID 2197679
- [Result] Visscher CM, Lobbezoo F, Naeije M. Comparison of algometry and palpation in the recognition of temporomandibular disorder pain complaints. J Orofac Pain. 2004 Summer;18(3):214-9. PMID 15509000
- [Result] Chesterton LS, Sim J, Wright CC, Foster NE. Interrater reliability of algometry in measuring pressure pain thresholds in healthy humans, using multiple raters. Clin J Pain. 2007 Nov-Dec;23(9):760-6. doi: 10.1097/AJP.0b013e318154b6ae. PMID 18075402
- [Result] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Result] Aydemir, Ö, Guvenir, T, Kuey, L, & Kultur, S. Validity and reliability of Turkish version of hospital anxiety and depression scale. Turk Psikiyatri Derg. 1997; 8(4); 280-287.
- [Result] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Result] Kocyigit H. Reliability and validity of the Turkish version of short form-36 (SF-36): a study in a group of patients will rheumatic diseases. Turk J Drugs Ther. 1999; 12; 102-106.
- [Result] Ohrbach R, Dworkin SF. Five-year outcomes in TMD: relationship of changes in pain to changes in physical and psychological variables. Pain. 1998 Feb;74(2-3):315-26. doi: 10.1016/s0304-3959(97)00194-2. PMID 9520246
- [Result] Gungormus Z, Erciyas K. Evaluation of the relationship between anxiety and depression and bruxism. J Int Med Res. 2009 Mar-Apr;37(2):547-50. doi: 10.1177/147323000903700231. PMID 19383250
- [Result] Manfredini D, Landi N, Romagnoli M, Bosco M. Psychic and occlusal factors in bruxers. Aust Dent J. 2004 Jun;49(2):84-9. doi: 10.1111/j.1834-7819.2004.tb00055.x. PMID 15293819
- [Result] Manfredini D, Winocur E, Guarda-Nardini L, Paesani D, Lobbezoo F. Epidemiology of bruxism in adults: a systematic review of the literature. J Orofac Pain. 2013 Spring;27(2):99-110. doi: 10.11607/jop.921. PMID 23630682
- [Result] Melis M, Abou-Atme YS. Prevalence of bruxism awareness in a Sardinian population. Cranio. 2003 Apr;21(2):144-51. doi: 10.1080/08869634.2003.11746243. PMID 12723861
- [Result] Pond LH, Barghi N, Barnwell GM. Occlusion and chewing side preference. J Prosthet Dent. 1986 Apr;55(4):498-500. doi: 10.1016/0022-3913(86)90186-1. No abstract available. PMID 3457182
- [Result] Santana-Mora U, Lopez-Cedrun J, Mora MJ, Otero XL, Santana-Penin U. Temporomandibular disorders: the habitual chewing side syndrome. PLoS One. 2013 Apr 8;8(4):e59980. doi: 10.1371/journal.pone.0059980. Print 2013. PMID 23593156
- [Result] Lee LT, Yeung RW, Wong MC, McMillan AS. Diagnostic sub-types, psychological distress and psychosocial dysfunction in southern Chinese people with temporomandibular disorders. J Oral Rehabil. 2008 Mar;35(3):184-90. doi: 10.1111/j.1365-2842.2007.01792.x. PMID 18254795
- [Result] Storm C, Wanman A. Temporomandibular disorders, headaches, and cervical pain among females in a Sami population. Acta Odontol Scand. 2006 Oct;64(5):319-25. doi: 10.1080/00016350600801915. PMID 16945899
- [Result] Resende CM, Alves AC, Coelho LT, Alchieri JC, Roncalli AG, Barbosa GA. Quality of life and general health in patients with temporomandibular disorders. Braz Oral Res. 2013 Mar-Apr;27(2):116-21. doi: 10.1590/s1806-83242013005000006. Epub 2013 Mar 1. PMID 23459771
- [Result] Wanman A. The relationship between muscle tenderness and craniomandibular disorders: a study of 35-year-olds from the general population. J Orofac Pain. 1995 Summer;9(3):235-43. PMID 8995923
- [Result] Almoznino G, Zini A, Zakuto A, Sharav Y, Haviv Y, Hadad A, Chweidan H, Yarom N, Benoliel R. Oral Health-Related Quality of Life in Patients with Temporomandibular Disorders. J Oral Facial Pain Headache. 2015 Summer;29(3):231-41. doi: 10.11607/ofph.1413. PMID 26244431
- [Result] Rener-Sitar K, Celebic A, Stipetic J, Marion L, Petricevic N, Zaletel-Kragelj L. Oral health related quality of life in Slovenian patients with craniomandibular disorders. Coll Antropol. 2008 Jun;32(2):513-7. PMID 18756903
- [Result] Vanderas AP, Menenakou M, Papagiannoulis L. Emotional stress and craniomandibular dysfunction in children. Cranio. 2001 Apr;19(2):123-9. doi: 10.1080/08869634.2001.11746161. PMID 11842863
- [Result] Moss RA, Adams HE. Physiological reactions to stress in subjects with and without myofascial pain dysfunction symptoms. J Oral Rehabil. 1984 May;11(3):219-32. doi: 10.1111/j.1365-2842.1984.tb00571.x. PMID 6588175
- [Result] Manfredini D, Landi N, Fantoni F, Segu M, Bosco M. Anxiety symptoms in clinically diagnosed bruxers. J Oral Rehabil. 2005 Aug;32(8):584-8. doi: 10.1111/j.1365-2842.2005.01462.x. PMID 16011637
- [Result] Kampe T, Edman G, Bader G, Tagdae T, Karlsson S. Personality traits in a group of subjects with long-standing bruxing behaviour. J Oral Rehabil. 1997 Aug;24(8):588-93. doi: 10.1046/j.1365-2842.1997.00541.x. PMID 9291252